CLINICAL TRIAL: NCT05566262
Title: An Investigator Initiated Open-label Study Evaluating the Efficacy and Tolerability of Application of Bodewell Products for the Treatment of Atopic Dermatitis
Brief Title: Bodewell Products for the Treatment of Atopic Dermatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Tiffany Mayo, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008755
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bodewell Treatment (Experimental): All patients will be treated with the active product, Bodewell. Bodewell will be applied topically twice a day to all active lesions.
  Interventions: Drug: Bodewell Calming Cream

INTERVENTIONS:
Drug: Bodewell Calming Cream — Bodewell is a non-prescription and contains 22 botanical ingredients in addition to colloidal oatmeal.

SUMMARY:
This study aims to examine the safety and efficacy of topical application of the Bodewell eczema products

ELIGIBILITY:
Inclusion Criteria:

1. In good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis. (NOTE: The definition of good health means a subject does not have uncontrolled significant co- morbid conditions).
2. 18 years of age or older
3. Able and willing to give written informed consent prior to any study procedures being conducted, and authorize the release and use of protected health information (PHI)
4. Willing to have photos taken of their skin
5. Diagnosis of chronic atopic dermatitis that has been present for at least 6 months prior to baseline
6. Atopic dermatitis involving at least 3-10 % of the patient's body surface area
7. Must have discontinued all systemic therapies for the treatment of atopic dermatitis at least 4 weeks or 5 half-lives, and biologics 6 months prior to baseline visit
8. Must have discontinued all topical therapies for the treatment of atopic dermatitis at least 2 weeks prior to baseline visit
9. Females of childbearing potential must use an approved birth control method while receiving treatment and for 28 days following the investigational product and there must be a documented negative pregnancy tests prior to initiating treatment. Approved birth control methods include hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring), intrauterine device, tubal ligation, partner vasectomy, or male or female condoms that are not made of natural materials PLUS a diaphragm with spermicide, cervical cap with spermicide, or a contraceptive sponge with spermicide.

   Females not of child bearing potential are defined as being at least 1 year postmenopausal or surgically sterile (bilateral tubal ligation, bilateral oophorectomy and/or hysterectomy).
10. 5 patients must be on a stable dose of systemic therapy for the last 6 months prior to screening visit
11. 5 patients must be skin of color

Exclusion Criteria:

1. Other than disease under study, any clinically significant (as determined by the Investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is currently uncontrolled
2. Any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he/she were to participate in the study
3. Prior history of suicide attempt at any time in the subject's life time prior to screening or randomization, or major psychiatric illness requiring hospitalization within the last 3 years
4. Pregnant or breast feeding
5. Active substance abuse or a history of substance abuse within 6 months prior to Screening
6. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer)
7. Prior treatment with the investigational product within 4 weeks prior to randomization
8. Unable to comply with the protocol (as defined by the Investigator; i.e. drug or alcohol abuse or history of noncompliance)
9. Any other dermatologic conditions that prohibit or confound the ability of the investigator to interpret skin findings.
10. Patients who will be unable to avoid the use of systemic steroids, excluding intranasal or inhaled steroids that will be permitted, for the duration of the trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Mean Percentage improvement in Patient Global Assessment (PGA) | Baseline to week 12
  Mean percentage improvement in the Patient Global Assessment from baseline to week 12. This assessment is a scale from 0 to 4. 0 means clear skin while 4 means severe disease.

SECONDARY OUTCOMES:
Percent improvement in Dermatology Life Quality Index (DLQI) | Baseline to week 12
  Percent improvement in Dermatology Life Quality Index (DLQI) from baseline to week 12. The DLQI consists of 10 questions, with each question being on a scale of 0 (clear) to 3 (more severe). The overall scoring scale is from 0 to 30. A higher score means a more severe outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Mayo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States